CLINICAL TRIAL: NCT06719232
Title: Evaluating the Efficacy and Patient Experience of Catheter-Free Intravesical Instillation: a Prospective Observational Study
Brief Title: Evaluating the Efficacy and Patient Experience of Catheter-Free Intravesical Instillation
Acronym: NOCATIN
Status: Recruiting | Type: Observational
Sponsor: Jahn Ferenc South Pest Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Béla Köves, Head Physician, Jahn Ferenc South Pest Teaching Hospital
Other Study IDs: NOCATIN
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Interstitial Cystitis; Recurrent Cystitis; Haemorrhagic Cystitis; Bladder Cancer; Bladder Disease; Intravesical Instillation; Bladder Pain Syndrome; Recurrent Urinary Tract Infections
Keywords: intravesical therapy; catheterization; recurrent urinary tract infection; IC/BPS; Interstitial Cystitis/Bladder Pain syndrome; Post-chemotherapy Cystitis; Post-Irradiation Cystitis; Intravesical instillation; UroDapter
MeSH Terms: conditions — Cystitis, Interstitial; Cystitis; Cystitis, Hemorrhagic; Urinary Bladder Neoplasms; Urinary Bladder Diseases; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Catheter-Free Intravesical Instillation Patients: This group consists of patients receiving catheter-free intravesical instillation treatments with a special syringe adapter, called UroDapter for any conditions, including interstitial cystitis/bladder pain syndrome (IC/BPS), recurrent urinary tract infections (UTIs), post-chemotherapy cystitis, post-radiation cystitis, and non-muscle invasive bladder cancer.
  Interventions: Device: Catheter-Free Intravesical Instillation with a special syringe adapter

INTERVENTIONS:
Device: Catheter-Free Intravesical Instillation with a special syringe adapter — The intervention involves catheter-free intravesical instillation using a specialized urological adapter. This device is attached to a syringe and inserted approximately 6-8 mm into the urethral opening, allowing the instillation solution to reach the bladder without the need for catheterization.

SUMMARY:
This study aims to evaluate a catheter-free method for delivering medications directly into the bladder, known as intravesical instillation, which is commonly used to treat conditions such as interstitial cystitis/bladder pain syndrome (IC/BPS), recurrent urinary tract infections, bladder cancer, and post-chemotherapy or post-radiation cystitis.

The study investigates whether this method, which eliminates the need for catheterization, reduces discomfort and complications while maintaining treatment effectiveness. By collecting data on patient experiences and outcomes, the study seeks to determine if this approach provides a safer and more comfortable alternative to traditional catheter-based treatments.

DETAILED DESCRIPTION:
Intravesical instillation, a method involving the direct administration of therapeutic agents into the bladder via a catheter, is widely used in the treatment of various urological conditions, including interstitial cystitis/bladder pain syndrome (IC/BPS), recurrent urinary tract infections (UTIs), post-chemotherapy and post-radiation cystitis, and non-muscle invasive bladder cancer. This approach allows high concentrations of medication to be delivered directly to the bladder without systemic exposure, thereby enhancing treatment efficacy while reducing the risk of systemic side effects.

A notable drawback of traditional intravesical treatments is the need for catheterization. However, catheter-free intravesical instillations have become possible with the use of a specialized urological adapter that requires only 6-8 mm insertion into the urethral opening (UroDapter). By relaxing the urethral sphincter, patients can facilitate the delivery of the instillation fluid into the bladder without a catheter. This method is painless, causes minimal discomfort, and significantly reduces the risk of urinary tract infections, urethral bleeding, and urethral strictures compared to catheter-based approaches. Catheter-free intravesical instillations have been performed in Hungarian outpatient urology settings since 2018.

This prospective observational study includes patients whose physicians recommended catheter-free bladder instillation therapy. The study aims to anonymously collect data on the treatment's effectiveness, patient experience and incidence of complications associated with the caheter-free approach, focusing on its application for IC/BPS, recurrent UTIs, post-chemotherapy and post-radiation cystitis, and bladder cancer. Findings will be instrumental in refining protocols for intravesical treatments and enhancing patient compliance and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged between 18 and 80 years.
* Patients for whom the treating physician has determined that intravesical instillation is necessary due to one of the following conditions:
* Interstitial cystitis/bladder pain syndrome (IC/BPS).
* Recurrent urinary tract infections (UTIs).
* Non-muscle invasive bladder cancer.
* Post-radiation cystitis.
* Post-chemotherapy cystitis.
* Negative urine culture within the last two weeks.
* Patients who provide verbal and written informed consent to participate in the study.

Exclusion Criteria:

* Urinary tract infection within the past month or currently active infection.
* Diagnosed bleeding disorders or recurrent macroscopic hematuria.
* Post-void residual urine volume greater than 100 ml.
* Mental condition that prevents reliable cooperation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients attending the participating centers. Study participants are individuals referred by their treating physicians for catheter-free intravesical instillation therapy based on their clinical needs.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient Discomfort During Catheter-Free Intravesical Instillation | Up to two weeks.
  Level of discomfort experienced by patients during catheter-free intravesical instillation treatments, measured using the Numerical Rating Scale (NRS) from 0 to 10

SECONDARY OUTCOMES:
Success Rate of Catheter-Free Instillation | During each instillation visit.
  Proportion of instillation procedures successfully completed as judged by the treating physician.
Incidence of Post-Treatment Urinary Tract Infections | Within 1-2 weeks following the last instillation.
  Occurrence of urinary tract infections post-treatment, confirmed by symptoms and positive urine culture.
Incidence of Urethral Bleeding | Within 2 weeks following the last instillation.
  Number of patients experiencing urethral bleeding during or after catheter-free intravesical instillation.
Patient Preference for Catheter-Free Instillation | Within 2 weeks following the last instillation.
  Percentage of patients preferring catheter-free intravesical instillation compared to previous catheter-based treatments (only in the sub-group of pts who had previous catheter-based treatments).
Incidence of Other Post-Treatment Complications | Within 2 weeks following the last instillation.
  Any additional complications related to catheter-free intravesical instillation, including pain or discomfort beyond expected levels.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tenke, Professor of Urology, Study Chair — South Pest Teaching Hospital
Locations (2):
- Hungary (2):
  - Military Hospital Medical Centre, Hungarian Defense Forces, Budapest
  - Jahn Ferenc South-Pest Hospital, Budapest

IPD SHARING:
Plan to Share IPD: Undecided